CLINICAL TRIAL: NCT06944158
Title: Antimicrobial Resistance (AMR) Knowledge, Attitudes, and Practices Among Healthcare Workers in Syria: Multicenter Cross Sectional Study
Brief Title: Antimicrobial Resistance (AMR) Study
Status: Recruiting | Type: Observational
Sponsor: University of Aleppo (Other)
Responsible Party: Principal Investigator, Ziad Al-Jarad, MD, University of Aleppo
Other Study IDs: AntibioticsResistance963
Record Dates: First submitted 2025-04-17; First posted 2025-04-25 (Actual); Last update posted 2025-04-25 (Actual); Status verified 2025-04

CONDITIONS: Anti-Microbial Resistance
Keywords: Antibiotics; Resistance; Knowledge

STUDY DESIGN:
Observational Model: Case-Crossover | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims to investigate the knowledge, attitudes and behaviours of the antibiotic resistance and prudent antibiotic use among healthcare workers in Syria

DETAILED DESCRIPTION:
This will be a multicenter cross-sectional study across the country.

The online questionnaire will be conducted in different governorates and published online through social media.

An online link to the web-based questionnaire will be developed using Google forms; it was self-designed based on questions used in previous similar studies[1]-[5].The questionnaire will take about 5-10 minutes to be completed by each participant.

The questionnaire consists of eight sections.

All participants fulfilling the inclusion criteria will be invited to participate. Snowball sampling will select the study participants with a confidence level of 95% and a margin of error of 5%. The lower limit of participants should be included is 200 healthcare workers.

The questionnaire will be pre-tested on a small sample of participants to confirm the practicability and clarity of questions to check the content. Observations of the pilot study will not be included in the final analysis.

Responses will be downloaded from Google form as an excel sheet, and data will be analyzed using SPSS version 28.

ELIGIBILITY:
Inclusion Criteria: We include healthcare workers, males or females aged 25 to over 65.

-

Exclusion Criteria: Participants who do not agree to fill the questionnaire, who do not agree to fill all requested questions, and who filled the questionnaire before.

-

Ages: 25 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The target population of this study is healthcare workers of both sexes (25-65 years old).
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2024-11-01 (Actual); Primary Completion 2025-06-01 (Estimated); Study Completion 2025-06 (Estimated)

PRIMARY OUTCOMES:
Knowledge, attitude and practice of health care workers (KAP) | 06/01/2025
  To evaluate the knowledge, attitudes, and practices (KAP) among healthcare workers of Antimicrobial resistance (AMR) in Syria

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, University of Aleppo, Aleppo, Syria